CLINICAL TRIAL: NCT01689324
Title: Immunogenicity and Safety of the Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine Adsorbed (SP306) as a Booster in Japanese Adolescents
Brief Title: Study of Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis Vaccine (ADACEL®) as a Booster in Adolescents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Td540; U1111-1124-7671 (Other: WHO)
Record Dates: First submitted 2012-09-17; First posted 2012-09-21 (Estimated); Results first posted 2014-02-21 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Pertussis; Tetanus; Diphtheria
Keywords: Pertussis; Tetanus; Diphtheria; Acellular pertussis; ADACEL®; Tdap vaccine
MeSH Terms: conditions — Whooping Cough; Tetanus; Diphtheria | interventions — adacel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental): Participants will receive a single booster dose of Tdap vaccine (ADACEL®) on Day 0.
  Interventions: Biological: (ADACEL®): Tetanus, Reduced Diphtheria Toxoid and Acellular Pertussis

INTERVENTIONS:
Biological: (ADACEL®): Tetanus, Reduced Diphtheria Toxoid and Acellular Pertussis — 0.5 mL, Intramuscular
  Other Names: ADACEL®; Tdap Vaccine

SUMMARY:
This study is designed to assess the immunogenicity and safety of tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine (ADACEL®, Tdap vaccine) as a booster dose in adolescents in Japan.

Primary Objective:

* To assess the immunogenicity of Tdap (SP306) when administered as a single dose in Japanese adolescents

Secondary Objective:

* To assess the safety of Tdap vaccine when administered as a single dose in Japanese adolescents.

DETAILED DESCRIPTION:
All participants will receive a single booster dose of Tdap vaccine (ADACEL®) on Day 0 and undergo immunogenicity assessment from blood samples provided prior to, and 28 days post-vaccination. Tolerability and safety will be monitored up to 28 days post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 11 or 12 years on the day of inclusion
* Informed consent form and assent form signed and dated by the parent(s) / legal representative and the subject respectively
* Completed childhood vaccination against diphtheria, pertussis and tetanus (i.e, received 4 doses of Japanese-produced tetanus toxoid, diphtheria toxoid and acellular pertussis vaccine absorbed [DTaP vaccine]), confirmed by checking immunization records and have not yet undergone additional adsorbed Diphtheria and Tetanus toxoid (DT) vaccination
* Able to attend all scheduled visits and to comply with all trial procedures
* For female subjects, either pre-menarchal, or post-menarchal with a negative urine pregnancy test.

Exclusion Criteria:

* Any conditions or diseases which, in the opinion of the investigator
* would pose a health risk to the subject
* or might interfere with the ability to participate fully in the study
* or might interfere with evaluation of the vaccine
* or would otherwise make participation inappropriate according to the investigator's clinical judgment
* History of diphtheria, tetanus, pertussis, confirmed either clinically, serologically, or microbiologically
* Known systemic hypersensitivity to any of the vaccine components or history of a life threatening reaction to a vaccine containing the same substances of the study vaccine
* Vaccination in the last 5 years against tetanus, diphtheria, and/or pertussis
* Known or suspected congenital immunodeficiency, or current / previous acquired immunodeficiency, or current / previous receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy, or current / previous (within the last 6 months) systemic corticosteroid therapy
* Participation in another clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 4 weeks preceding the trial inclusion
* Planned participation in another clinical trial during the present trial period
* Receipt of blood or blood-derived products in the past 3 months, that might interfere with assessment of the immune response
* Receipt of any vaccine within the 4 weeks preceding the trial vaccination, except for influenza vaccination, which may be received at least 2 weeks before the study vaccine
* Planned receipt of any vaccine during the trial period
* Clinical or known serological evidence of systemic illness including Hepatitis B, Hepatitis C and/or Human Immunodeficiency Virus (HIV) infection
* At high risk for diphtheria, tetanus or pertussis infection during the trial
* Known pregnancy, or a positive urine pregnancy test
* Currently breastfeeding a child
* Known thrombocytopenia, contraindicating intramuscular (IM) vaccination, or a history of thrombocytopenia
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination
* History of acute disseminated encephalomyelitis, encephalopathy, Guillain-Barré Syndrome (GBS), or autoimmune disease
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction that might interfere with the ability to comply with trial procedures
* Identified as an employee of an Investigator, a study center, a study-affiliated vendor, or the Sponsor, with direct or indirect involvement in the proposed study or other studies under the direction of that Investigator or study center; or identified as a spouse or child (whether natural or adopted) of such an employee.

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur K.K
Locations (3):
- Japan (3):
  - Aichi
  - Ibaraki
  - Nagano

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were enrolled from 12 September through 14 October 2012 in 3 clinic centers in Japan.
Pre-assignment Details: A total of 43 participants that met all the inclusion criteria but none of the exclusion criteria were enrolled and vaccinated in the study.
Groups:
- Study Group: Participants received a single booster dose of Tetanus Toxoid, Reduced Diphtheria Toxoid and Acellular Pertussis vaccine (Tdap vaccine; ADACEL®) on Day 0.
Period: Overall Study
Arm/Group | Study Group
Started | 43
Completed | 43
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Study Group
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 43
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.4 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 20
Region of Enrollment [Number; unit: Participants]
  Japan | 43

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Seroprotection Against Diphtheria and Tetanus Antigens Following Vaccination With ADACEL®
Description: Seroprotection was defined as the percentage of participants with antibody concentration of ≥0.1 IU/mL, post-vaccination.
Time Frame: Day 28 post-vaccination
Population: Seroprotection to diphtheria and tetanus antigens were determined in the Immunology Analysis Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Study Group
Number analyzed (Participants) | 43
Percentage of Participants
  Diphtheria | 100
  Tetanus | 100

2. Primary Outcome: Percentage of Participants With Booster Response to Diphtheria and Tetanus Antigens Following Vaccination With ADACEL®
Description: Diphtheria booster response was defined as a ≥ 4-fold rise in pre- to post-vaccination antitoxin concentration in a subject with a pre-vaccination antitoxin concentration ≤ 2.56 IU/mL; or a ≥ 2-fold rise in a subject with a pre-vaccination antitoxin concentration > 2.56 IU/mL.
  Tetanus booster response was defined as a ≥ 4-fold rise in pre- to post- vaccination antitoxin concentration in a subject with a pre-vaccination antitoxin concentration ≤ 2.7 IU/mL; or a ≥ 2-fold rise in a subject with a pre-vaccination antitoxin concentration > 2.7 IU/mL.
Time Frame: Day 28 post-vaccination
Population: Booster response to diphtheria and tetanus antigens were determined in the Immunology Analysis Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Study Group
Number analyzed (Participants) | 43
Percentage of Participants
  Diphtheria | 98
  Tetanus | 100

3. Primary Outcome: Percentage of Participants With Booster Response to Pertussis Antigens, Pertussis Toxoid and Filamentous Hemagglutinin Following Vaccination With ADACEL®
Description: Booster responses were defined as: Pre-vaccination antibody concentrations less than the lower limit of quantitation (LLOQ) and a post-vaccination levels ≥ 4x LLOQ; or Pre-vaccination antibody concentrations ≥ LLOQ but < 4x LLOQ, and a 4-fold rise (i.e., post-/pre-vaccination ≥ 4), or Pre-vaccination antibody concentrations ≥ 4x LLOQ and a 2-fold rise (i.e., post-/pre-vaccination ≥ 2)
Time Frame: Day 28 post-vaccination
Population: Booster response to pertussis antigens were determined in the Immunology Analysis Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Study Group
Number analyzed (Participants) | 43
Percentage of Participants
  Pertussis toxoid | 63
  Filamentous hemagglutinin | 88

4. Other Pre Specified Outcome: Percentage of Participants With Seroprotection Against Diphtheria and Tetanus Antigens Pre-vaccination With ADACEL®
Description: Seroprotection was defined as the percentage of participants with antibody concentration of ≥0.1 IU/mL.
Time Frame: Day 0 pre-vaccination
Population: Pre-vaccination seroprotection to diphtheria and tetanus antigens were determined in the Immunology Analysis Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Study Group
Number analyzed (Participants) | 43
Percentage of Participants
  Diphtheria | 63
  Tetanus | 91

5. Other Pre Specified Outcome: Percentage of Participants With Seroprotection Against Diphtheria and Tetanus Pre-vaccination and Post-vaccination With ADACEL®
Description: Seroprotection was defined as the percentage of participants with antibody concentration of ≥0.01 IU/mL.
Time Frame: Day 0 (pre-vaccination) and day 28 post-vaccination
Population: Pre- and post-vaccination seroprotection to diphtheria and tetanus antigens were determined in the Immunology Analysis Set.
Measure: Number; unit: Percentage of Participants
Arm/Group | Study Group
Number analyzed (Participants) | 43
Percentage of Participants
  Diphtheria (Pre-vaccination) | 100
  Diphtheria (Post-vaccination) | 100
  Tetanus (Pre-vaccination) | 100
  Tetanus (Post-vaccination) | 100

6. Other Pre Specified Outcome: Percentage of Participants With Seroprotection Against Diphtheria and Tetanus Antigens Pre-vaccination and Post-vaccination With ADACEL®
Description: Seroprotection was defined as the percentage of participants with antibody concentration of ≥1.0 IU/mL.
Time Frame: Day 0 (pre-vaccination) and day 28 post-vaccination
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Study Group
Number analyzed (Participants) | 43
Percentage of Participants
  Diphtheria (Pre-vaccination) | 12
  Diphtheria (Post-vaccination) | 100
  Tetanus (Pre-vaccination) | 30
  Tetanus (Post-vaccination) | 100

7. Other Pre Specified Outcome: Geometric Mean Concentrations With Respect to Diphtheria and Tetanus Antibodies Pre- and Post-vaccination With ADACEL®
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Pre and post vaccination geometric mean concentrations to Diphtheria and Tetanus antigens were determined in the Immunology Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Study Group
Number analyzed (Participants) | 43
Titers
  Diphtheria (Pre-vaccination) | 0.22 [0.14 to 0.35]
  Diphtheria (Post-vaccination) | 8.58 [6.76 to 10.88]
  Tetanus (Pre-vaccination) | 0.46 [0.33 to 0.64]
  Tetanus (Post-vaccination) | 37.80 [30.16 to 47.38]

8. Other Pre Specified Outcome: Geometric Mean Concentrations With Respect to Pertussis Antibodies Pre- and Post-vaccination With ADACEL®
Time Frame: Day 0 (pre-vaccination) and Day 28 post-vaccination
Population: Pre and post vaccination geometric mean concentrations to pertussis antibodies were determined in the Immunology Analysis Set
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Study Group
Number analyzed (Participants) | 43
Titers
  Pertussis toxoid (pre-vaccination) | 12.21 [7.82 to 19.05]
  Pertussis toxoid (post-vaccination) | 46.92 [33.65 to 65.42]
  Filamentous hemagglutinin (pre-vaccination) | 34.79 [23.47 to 51.57]
  Filamentous hemagglutinin (post-vaccination) | 204.00 [164.26 to 253.36]
  Pertactin (pre-vaccination) | 10.64 [6.28 to 18.03]
  Pertactin (post-vaccination) | 272.82 [197.63 to 376.62]
  Fimbriae types 2 and 3 (pre-vaccination) | 7.78 [5.42 to 11.17]
  Fimbriae types 2 and 3 (post-vaccination) | 748.28 [443.23 to 1263.27]

9. Other Pre Specified Outcome: Percentage of Participants With Booster Response to Pertussis Antigens, Pertactin and Fimbriae Following Vaccination With ADACEL®
Description: as for outcome 3
Time Frame: Day 28 post-vaccination
Population: Booster response to pertussis antigens were determined in the Immunology Analysis Set
Measure: Number; unit: Percentage of Participants
Arm/Group | Study Group
Number analyzed (Participants) | 43
Percentage of Participants
  Pertactin | 93
  Fimbriae Types 2 and 3 | 98

10. Other Pre Specified Outcome: Number of Participants Reporting Solicited Injection-site and Systemic Reactions Following Vaccination With ADACEL®
Description: Solicited injection-site reactions: Pain, Redness, and Swelling. Grade 3: Pain, Significant, prevents daily activity; Redness and Swelling, >100 mm.
  Solicited systemic reactions: Fever (Temperature); Headache, Malaise, and Myalgia. Grade 3: Fever, ≥ 39°C; Headache, Malaise and Myalgia, Significant, prevents daily activity.
Time Frame: Day 0 up to Day 7 post-vaccination
Population: Solicited injection site and systemic reactions were assessed in the Safety Analysis Set
Measure: Number; unit: Participants
Arm/Group | Study Group
Number analyzed (Participants) | 43
Participants
  Solicited injection site Pain | 37
  Grade 3 solicited injection site Pain | 0
  Solicited injection site Erythema | 9
  Grade 3 solicited injection site Erythema | 0
  Solicited injection site Swelling | 12
  Grade 3 solicited injection site Swelling | 1
  Fever | 9
  Grade 3 Fever | 1
  Headache | 8
  Grade 3 Headache | 0
  Malaise | 11
  Grade 3 Malaise | 0
  Myalgia | 17
  Grade 3 Myalgia | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from Day 0 (post-vaccination) up to 1 month post-vaccination
Groups:
- Study Group: Participants received a single booster dose of Tdap vaccine on Day 0.
Arm/Group | Study Group
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 39/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=43)
Solicited injection site Pain (General disorders) | 37 (37)
Solicited injection site Erythema (General disorders) | 9 (9)
Solicited injection site Swelling (General disorders) | 12 (12)
Fever (General disorders) | 9 (9)
Malaise (General disorders) | 11 (11)
Myalgia (General disorders) | 17 (17)
Nasopharyngitis (Infections and infestations) | 7 (9)
Headache (Nervous system disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.